CLINICAL TRIAL: NCT03192878
Title: A Prospective Observational Study of Infliximab Biosimilar in the Treatment of Takayasu's Arteritis Resistant to Corticosteroids and Conventional Immune-suppressive Treatments
Brief Title: Infliximab Biosimilar in Takayasu's Arteritis
Acronym: TAKASIM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Lorenzo Dagna, Head, Unit of Immunology, Rheumatology, Allergy and Rare Diseases, Ospedale San Raffaele
Other Study IDs: TakaSim
Record Dates: First submitted 2017-05-09; First posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Takayasu Arteritis
Keywords: infliximab; biosimilars; treatment
MeSH Terms: conditions — Takayasu Arteritis | interventions — Infliximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Naive patients: Patients with corticosteroid- and/or traditional immunosuppressive drug-resistant Takayasu's arteritis with indication of initiating therapy with anti-TNF-alpha
  Interventions: Drug: Infliximab
- Switch patients: Patients with Takayasu's arteritis already in therapy with infliximab originator (Remicade) in whom the originator therapy will be replaced with infliximab biosimilar therapy
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — infliximab biosimilar

SUMMARY:
Takayasu arteritis (TA) is a chronic inflammatory disease affecting large and medium caliber arteries, particularly the aortic arch and its main branches. Clinical manifestations are caused by the marked thickening of the wall of the involved vessels, resulting in lumen narrowing and ischemia of the tributary districts. Therapy is based on the use of corticosteroids, immunosuppressants, and biologic drugs including infliximab, a monoclonal antibody blocking tissue necrosis factor (TNF)-alpha. Biosimilar infliximab is commercially available and used in the treatment of various immune-mediated conditions. There are currently no data on the efficacy and safety of biosimilar infliximab in the treatment of TA.

The investigators propose this monocentric, observational, prospective, open label study to evaluate the efficacy and safety of biosimilar infliximab in the treatment of 30 patients with TA. Specifically, the study will include: I) TA patients refractory to treatment with corticosteroid and/or immmunosuppressive therapy, not previously treated with infliximab; II) TA patients already receiving treatment with originator infliximab.

Biosimilar infliximab will be administered at dosages usually employed in the treatment of TA. Specifically, patients not previously treated with the originator drug will receive biosimilar infliximab intravenously at a dose of 5 mg/Kg at time 0, at week 2, at week 4; thereafter, treatment will be administered every 4-6 weeks at a dose of 5-10 mg/kg based on clinical judgement. In patients previously treated with the originator drug, biosimilar infliximab will be administered at the same dosages.

To evaluate the efficacy of therapy, changes in clinical manifestations, laboratory examinations, and imaging findings including angio-magnetic resonance imaging (MRI) of thoracic and abdominal vessels and total body PET/CT scan will be evaluate at time 0 as well as 6 and 12 months following treatment initiation. In order to evaluate the safety of the study treatment, the investigators will stringently evaluate possible side effects of treatment, including infusion reactions, changes in laboratory tests, infection, cancer, autoimmune manifestations, neurological and cardiovascular symptoms.

The total duration of follow up for each patient will be 52 weeks from enrolment.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years;
* negative pregnancy test;
* use of a reliable contraceptive method by all potentially fertile patients during the study and for the six months following the end of therapy;
* diagnosis of TA according to the Classification criteria of the American College of Rheumatology 1990;
* Multifocal vascular aortic and arterial involvement as evaluated by imaging examinations (angiography / angio-MRI / vascular ecocolordoppler / PET);
* failure to respond to corticosteroid therapy after 6-8 weeks of prednisone therapy at a dose of 1 mg / Kg per day, or impossibility to reduce the dose of prednisone to 0.5 mg / Kg within 3 months of initiation of therapy and to less than 0.2 mg / kg per day within 6 months of initiation of therapy (may also include patients who, despite receiving combination therapy with prednisone and cyclophosphamide, azathioprine, methotrexate, cyclosporin A, mycophenolate mofetil, leflunomide and rapamycin for at least 3 months, could not reduce the prednisone dose to 0.5 mg / Kg per day within 3 months of initiation of therapy, or to less than 0.2 mg / kg per day within 6 months of initiation of therapy);
* ongoing anti-TNF-alpha treatment with originator infliximab (inclusion criterion for the switch arm).

Exclusion Criteria:

* history of lymphoproliferative disease or solid neoplasm in the last 5 years, with the exception of successfully treated and completely resolved squamous cell skin carcinoma;
* history of uncontrolled diabetes, unstable cardiac ischaemia, congestive heart failure (NYHA class III and IV), active intestinal inflammatory disease, active peptic ulcer, recent stroke (within 3 months) and any other pathological conditions that, according to the treating physician, could expose the subject to the risk of adverse events;
* serological tests for hepatitis B or C indicating an active infection;
* history of HIV infection;
* chronic infection, or severe infections requiring hospitalization or intravenous antibiotic treatment within 30 days prior to inclusion in the study, or requiring treatment with oral antibiotics within 14 days prior to enrollment;
* ongoing pregnancy or lactation;
* history of drug or alcohol abuse;
* Previous diagnosis or signs of demyelinating disease of the central nervous system;
* history of active tuberculosis, histoplasmosis or listeriosis;
* previous infection with M. tuberculosis (as documented by chest x-rays and / or positive quantiferon test), in which case patients will only be enrolled after initiating prophylactic therapy according to current guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We anticipate to include about 30 patients with Takayasu's arteritis (TA). Specifically, the study will include:
  I) TA patients refractory to treatment with corticosteroid and/or immmunosuppressive therapy, not previously treated with infliximab (the naive arm).
  II) TA patients refractory to treatment with corticosteroid and/or immmunosuppressive therapy, already receiving treatment with originator infliximab (the switch arm).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients with active disease at month 6 | 6 months of treatment
  Disease will be defined active when new vascular lesion(s) (aneurysms, stenoses or occlusions, new arterial-wall irregularities) will be detected in arteries (aorta, innominate, subclavian, axillary, common and internal carotid, vertebral, superior and inferior mesenteric, renal, common iliac, and celiac axis) by MRI angiography or when increased arterial glucose uptake will be detected by FDG-PET scanning. Disease will also be defined active if at least 2 of the following will be present: 1) new onset of carotodynia or pain over large vessels, 2) transient ischemic episodes not attributable to other factors, 3) new bruit or new asymmetry in pulses or blood pressure determination, 4) ischemic symptoms (including new-onset claudication), and 5) fever in absence of infection
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 12 months of treatment
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 at month 12

SECONDARY OUTCOMES:
Number of patients with active disease at month 12 | 12 months of treatment
  Disease will be defined active when new vascular lesion(s) (aneurysms, stenoses or occlusions, new arterial-wall irregularities) will be detected in arteries (aorta, innominate, subclavian, axillary, common and internal carotid, vertebral, superior and inferior mesenteric, renal, common iliac, and celiac axis) by MRI angiography or when increased arterial glucose uptake will be detected by FDG-PET scanning. Disease will also be defined active if at least 2 of the following will be present: 1) new onset of carotodynia or pain over large vessels, 2) transient ischemic episodes not attributable to other factors, 3) new bruit or new asymmetry in pulses or blood pressure determination, 4) ischemic symptoms (including new-onset claudication), and 5) fever in absence of infection
Impact of the treatment on quality of life as assessed by the HAQ questionnaire | 6 months of treatment
  We will evaluate the changes from baseline in the HAQ questionnaires at month 6
Impact of the treatment on quality of life as assessed by the HAQ questionnaire | 12 months of treatment
  We will evaluate the changes from baseline in the HAQ questionnaires at month 12
Impact of the treatment on quality of life as assessed by the SF36 questionnaire | 6 months of treatment
  We will evaluate the changes from baseline in the SF36 questionnaire at month 6
Impact of the treatment on quality of life as assessed by the SF36 questionnaire | 12 months of treatment
  We will evaluate the changes from baseline in the SF36 questionnaire at month 12
Changes in the serum levels of TNF-alpha and anti-infliximab antibodies before and upon treatment with biosimilar infliximab. | 6 months of treatment
  Levels of TNF-alpha and anti-infliximab antibodies will be determined by an immunoenzymatic assay and compared to reference ranges provided by the manufacturer. Serum levels of TNFα are expected to decrease upon treatment with biosimilar infliximab; generation of anti-infliximab antibodies may occur in some patients and may be associated with reduced treatment efficacy.
Changes in the serum levels of TNF-alpha and anti-infliximab antibodies before and upon treatment with biosimilar infliximab. | 12 months of treatment
  Levels of TNF-alpha and anti-infliximab antibodies will be determined by an immunoenzymatic assay and compared to reference ranges provided by the manufacturer. Serum levels of TNFα are expected to decrease upon treatment with biosimilar infliximab; generation of anti-infliximab antibodies may occur in some patients and may be associated with reduced treatment efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Dagna, MD, Principal Investigator — IRCCS H San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided